CLINICAL TRIAL: NCT05679544
Title: Biological Signatures (Proteomics, Metabolomics and Genotoxicity) Associated With Occupational Exposure to PAH Mixtures and Relation With Exposure Biomarkers: Support for the Derivation of Biological Limit Values
Brief Title: Biological Signatures Resulting From Occupational Exposure to Complex Mixtures of PAHs
Acronym: PAH-ProMetGen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38RC22.0219; 2022-A01590-43 (Other: IDRCB)
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Disturbance; Protein Deficiency; Genotoxicity
Keywords: polycyclic aromatic hydrocarbons; metabolism; mixtures; occupational exposure; genotoxicity
MeSH Terms: conditions — Protein Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects occupationally exposed to PAHs (Experimental)
  Interventions: Biological: Characterization of early biological effects following exposure to PAHs

INTERVENTIONS:
Biological: Characterization of early biological effects following exposure to PAHs — Biological samples collected in period of exposure and after holidays

SUMMARY:
This research project aims at better understanding the early biological effects resulting from occupational exposure to complex Polycyclic Aromatic Hydrocarbon (PAH) mixtures.

Current biomarkers used as part of biomonitoring campaigns are biomarkers of exposure, not numerous and poorly related to health effects.

The aim of this study is thus to improve our understanding of biological consequences of such exposures, both in terms of proteins deregulation, metabolism deregulation and genotoxicity.

DETAILED DESCRIPTION:
PAHs are ubiquitous pollutants inducing several diseases, among which cancer is the most significant endpoint, with increased incidences of lung, skin, and bladder cancers. PAHs induce genotoxic effects (sister chromatids exchange, micronuclei, DNA damage) but require metabolic activation in humans as indirect-acting carcinogens. Thus, the knowledge of metabolic pathways involved following PAH exposure is critical for understanding and preventing cancer risks. Besides, exposure to PAHs is assumed to induce other adverse health effects (diabetes, inflammation, infertility, cardiovascular disease). Unfortunately, early disease-related biomarkers are still largely unknown and our comprehension about the mechanisms involved is still limited. The rare existing biological limit values either refer to not carcinogenic PAH (pyrene) or detoxification pathways (3-OHBaP for BaP), although new biomarkers reflecting the genotoxic pathway of BaP (TetraolBaP) are now available. There is thus a need for identifying more relevant biomarkers of exposure / effect, and for a better understanding of the biological consequences resulting from PAH exposures as well as the associated metabolic pathways involved.

The objectives of the project are :

* To better understand and characterize molecular, metabolic and genotoxic impacts resulting from exposure to PAHs and to link such impacts with biological levels of various PAH metabolites,
* To study the influence of BaP metabolism (genotoxic versus detoxication pathway) on the differential expression of metabolites / proteins and on genotoxicity endpoints in order to get relevant data for deriving new biological limit values,
* To elucidate the associations between omics deregulations due to PAH exposures and activated metabolic pathways, in order to define candidate effect biomarkers for human biomonitoring.

The originalities of the project are the following. First, this is a human study performed in real occupational settings on workers exposed to representative PAH mixtures. It is a multidisciplinary approach simultaneously combining up-to-date biomonitoring, omics and cytogenetics analyses, that will give insight into a comprehensive view of metabolic reactions and protein expressions following occupational exposure to PAH mixtures, and allow the identification of the biological processes involved. Carcinogenic BaP metabolites (Tetraol-BaP and 3-OHBaP) will be simultaneously analyzed in order to compare the two main metabolic pathways of BaP.

The main steps of the projects will be :

* Recruitment of 100 workers differentially exposed to PAH mixtures sampled across two time periods (after weeks of exposure and following 3 weeks without occupational exposure),
* Recording of relevant data (work characteristics, jobs / tasks, working experience, number of years of exposure, smoking habits, nutritional intake, co-morbidity),
* Toxicological analyses (LC-Fluorescence and GC-MS-MS) of urinary metabolites of several gaseous and particulate PAHs (Naphtalene, Fluorene, Phenanthrene, Pyrene, BaP, BeP, Chrysene, Benzo(b)Fluoranthene, Benzo(k)Fluoranthene, Benzo(a)Anthracene),
* Proteomics analyses on blood samples through an enrichment approach for a bottom-up label free quantitative proteomic analysis based LC-HR-MS. Deregulated proteins (DEP) will be identified and the associated protein signature. A gene ontology (GO) analysis will define the groups of biological processes involved,
* Untargeted Metabolomics analyses on blood samples in UHPLC-HR-MS, with unsupervised statistical analyses (Principal Component Analysis, Logistic Regressions), identification of relevant metabolites by their comparison to the Human Metabolome database, and advanced molecular networking / spectral library search of LC-MSMS data,
* Micronuclei (MN) in buccal cells through the harvesting of buccal cells using a cytobrush, transfer to the lab in a buffer, fixing and staining, automatic counting under fluorescent light.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18 years or more
* Subjects occupationally exposed to PAHs since more than 3 months
* Having signed the informed consent
* recruited by the occupational health service

Exclusion Criteria:

* Obesity (BMI>30)
* Subjects suffering cancers or metabolic diseases (diabetes, dyslipidemia, amino-acid diseases, renal or hepatic impairment) at the onset of the study.
* Subjects taking medications related to the above diseases at the onset of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Deregulation of blood proteins expression due to exposure to PAHs | up to 6 months between both periods of study
  Number of proteins up or down regulated in period of exposure versus after holidays
Deregulation of blood metabolites expression due to exposure to PAHs | up to 6 months between both periods of study
  Number of metabolites up or down regulated in period of exposure versus after holidays
Frequency of micronuclei measured due to exposure to PAHs | up to 6 months between both periods of study
  Frequency of cells containing micronuclei in period of exposure versus after holidays

CONTACTS AND LOCATIONS:
Overall Officials: Renaud PERSOONS, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No